CLINICAL TRIAL: NCT05087758
Title: An Open-Label Trial to Assess the Clinical Effectiveness of Matrion™ Decellularized Placental Membrane in Subjects With Diabetic Foot Ulcers
Brief Title: Matrion™ Decellularized Placental Membrane in Subjects With Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeNet Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-21-001
Record Dates: First submitted 2021-10-10; First posted 2021-10-21 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Foot; Lower Extremity Wound
Keywords: diabetic foot ulcer; placental membrane; lower extremity wound; decellularized placental membrane
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: The study is a multicenter, randomized, controlled, open-label trial designed to evaluate the safety and efficacy of Matrion on the wound healing rate of diabetic foot ulcers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Matrion decellularized placental membrane (Experimental): Matrion placental membrane graft will be use to treat subjects diagnosed with a diabetic foot ulcer.
  Interventions: Other: Matrion
- Conventional Care Wound Management (Active Comparator): Currently accepted standard of care wound management including Conventional care dressings will be utilized in subjects with a diabetic foot ulcer diagnosis.
  Interventions: Other: Conventional Care Wound Management

INTERVENTIONS:
Other: Matrion — Decellularized placental membrane applied to Wagner 1 and 2 diabetic foot ulcers
  Arms: Matrion decellularized placental membrane
Other: Conventional Care Wound Management — Advanced wound care with debridement and dressings
  Arms: Conventional Care Wound Management

SUMMARY:
In this study, a novel placental membrane product Matrion™ (LifeNet Health, Inc., Virginia Beach, VA) will be used as a treatment for subjects with diabetic foot ulcers. Matrion is composed of placental membrane derived from donated human birth tissue containing both the innermost amniotic layer and the outermost chorionic layer, inclusive of the trophoblast layer. Matrion is minimally processed and disinfected using a proprietary decellularization technology and terminally sterilized that safely renders the placental membrane acellular and sterile for its intended surgical applications.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible to participate in the study, a subject must meet the inclusion criteria listed below:

1. Be male or female, between 21 and 80 years of age at the time of consent
2. For subjects with a diagnosis of Type I or Type II diabetes as defined by the American Diabetes Association, have been on a stable anti-diabetic treatment for at least 30 days before the baseline visit
3. Have a full-thickness wound of the lower extremity
4. Have a single target ulcer
5. Have a wound with an area greater than or equal to 1 cm2 and less than 25 cm2 and a depth less than or equal to 9 mm
6. Have a diabetic foot ulcer that has been present for at least 30 days with a Wagner Classification Grade 1 or 2:

   * Grade 1: superficial diabetic ulcer including the full skin thickness but not underlying tissue
   * Grade 2: ulcer extension involving ligament, tendon, joint capsule, or fascia, without presence of abscess of osteomyelitis
7. Have an absence of infection based on Infectious Disease Society of America criteria
8. Have an adequate circulation to the affected lower extremity, defined as at least one these criteria:

   * Transcutaneous oxygen measurement at the dorsum of the foot greater or equal to 30 mmHg
   * Ankle-brachial index (ABI) greater than 0.75
   * At least biphasic Doppler arterial waveforms at the dorsalis pedis and posterior tibial arteries
9. Have the ability to comply with off-loading (if required for specific wound) and dressing change requirements
10. Have the ability to understand the requirements of the study, have provided written informed consent as evidenced by signature on an informed consent form (ICF) approved by an institutional review board (IRB), and agree to abide by the study restrictions and return to the site for the required assessments
11. Have provided written authorization for use and disclosure of protected health information
12. Have a life expectancy of greater than 6 months

Exclusion Criteria:

To be eligible for entry into the study, the subject must not meet any of the exclusion criteria listed below:

1. Be pregnant or lactating
2. Have a wound that decreased in size ≥50% between the Screening and Baseline Visits
3. Have circulating hemoglobin A1c exceeding 12% within 90 days of the Screening Visit
4. Have serum creatinine concentrations of 3.0 mg/dL or greater within 30 days prior to screening
5. Have a sensitivity to any of the following antibiotics: Lincomycin, Polymyxin B Sulfate, and/or Vancomycin
6. Have a sensitivity to N-Lauroyl Sarcosinate, and/or Benzonase® or Denarase®
7. Have the wound treated with biomedical or topical growth factors within the previous 30 days before the screening visit
8. Need for any additional concomitant dressing material other than the ones approved for this study
9. Have clinical signs of an infection at the study ulcer site
10. Have the inability to tolerate off-loading (a surgical shoe, removable cast walker or a total contact cast)
11. Have a known or suspected disease of the immune system
12. Have an active or untreated malignancy or active, uncontrolled connective tissue disease
13. Had a treatment with immunosuppressive or chemotherapeutic agents, radiotherapy or systemic corticosteroids less than 30 days before the baseline visit
14. Have presence of necrosis, purulence, or sinus tracts that cannot be removed by debridement
15. Has undergone a revascularization procedure aimed at increasing blood flow in the treatment target limb less than 4 weeks before the baseline visit
16. Have serum aspartate aminotransferase, alanine aminotransferase, or alkaline phosphatase levels greater than three times the normal upper limit within 30 days prior to screening
17. Have evidence of active Charcot disease
18. Have undergone treatment with a living skin equivalent within the last 4 weeks before screening
19. Have ongoing evidence of peripheral vascular disease, including greater than one nonpalpable pulse on either foot
20. Have the presence of any condition that in the opinion of the investigator places the subject at undue risk or potentially jeopardizes the quality of the data to be generated

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Wound Healing | 12 weeks
  Proportion of chronic DFUs that have achieved complete wound closure

SECONDARY OUTCOMES:
Speed of Wound Closure | 12 weeks
  Time to wound closure measured from the baseline visit to the termination visit
Wound Area | 12 weeks
  Change in wound area over time
Infection | 12 weeks
  Rate of wound infection
Reoccurrence | 6 months post termination visit
  Rate of reoccurrence of wound post treatment
Grafts Used | 12 weeks
  Average number of Matrion grafts used per subject
Incidence of Treatment Emergent Adverse Events | 12 weeks
  Collection of adverse events, including changes in vital signs, ABI, and physical exams

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Compass Medical Research Center, LLC, Tucson, Arizona
  - Center for Clinical Research, INC, Carmichael, California
  - Limb Preservation Platform, INC, Fresno, California
  - ILD Research Center, San Diego, California
  - Center for Clinical Research, INC, San Francisco, California
  - Doctors Research Network, Miami, Florida
  - Albuquerque Associated Podiatrists, Albuquerque, New Mexico
  - Purvis-Moyer Foot and Ankle Center, Rocky Mount, North Carolina

IPD SHARING:
Plan to Share IPD: No